CLINICAL TRIAL: NCT02593760
Title: A Phase IB/III, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Vismodegib in Combination With Ruxolitinib Versus Placebo and Ruxolitinib in Patients With Intermediate- or High-Risk Myelofibrosis
Brief Title: A Study to Evaluate the Efficacy and Safety of Vismodegib in Combination With Ruxolitinib for the Treatment of Intermediate- or High-Risk Myelofibrosis (MF)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WO29806; 2015-001620-33 (EudraCT Number)
Record Dates: First submitted 2015-10-29; First posted 2015-11-02 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Myelofibrosis
MeSH Terms: conditions — Primary Myelofibrosis | interventions — ruxolitinib; HhAntag691

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo + Ruxolitinib (Active Comparator): Participants will receive placebo (PO QD) in combination with ruxolitinib (dose will depend on the participant's baseline platelet count) for up to 48 weeks.
  Interventions: Other: Placebo; Drug: Ruxolitinib
- Vismodegib + Ruxolitinib (Experimental): Participants will receive vismodegib (150 mg PO QD) in combination with ruxolitinib (dose will depend on the participant's baseline platelet count) for up to 48 weeks.
  Interventions: Drug: Ruxolitinib; Drug: Vismodegib

INTERVENTIONS:
Other: Placebo — Placebo will be administered PO QD for up to 48 weeks.
  Arms: Placebo + Ruxolitinib
Drug: Ruxolitinib — Ruxolitinib will be administered PO BID at a starting dose depending on the participants's baseline platelet count for up to 48 weeks.
Drug: Vismodegib — Vismodegib will be administered at a dose of 150 mg PO QD for up to 48 weeks.
  Other Names: Erivedge
  Arms: Vismodegib + Ruxolitinib

SUMMARY:
This multicenter, randomized, double-blind, placebo-controlled study will evaluate the efficacy and safety of vismodegib plus (+) ruxolitinib versus placebo + ruxolitinib in participants with intermediate- or high-risk MF. The study will be divided into 2 components. The Phase Ib portion of the study consists of participants receiving open-label vismodegib (150 milligrams [mg] orally [PO] once daily [QD]) + ruxolitinib (PO twice daily [BID]). A safety assessment will be performed after the first 10 participants have been treated for 6 weeks. An analysis for efficacy and safety is planned in the first 10 participants at Week 24. There will be a hold on participant screening and enrollment during this assessment. Another 10 participants may be enrolled, thereafter, to further assess efficacy and safety (at Week 24) before the initiation of the Phase III randomization portion of the study. Similarly, there will be another hold on participant screening and enrollment during this assessment. The participants enrolled in the Phase Ib portion of the study will continue to receive vismodegib (150 mg PO QD) + ruxolitinib (PO BID) for up to 48 weeks, if clinical benefit is observed after 24 weeks. The Phase III randomized, double-blind portion of the study will enroll approximately 84 participants. Participants will be randomly assigned in a 1:1 ratio (double blind) to receive either vismodegib (150 mg PO QD) + ruxolitinib (PO BID) or placebo (PO QD) + ruxolitinib (PO BID) for up to 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed diagnosis of primary MF, post-polycythemia vera MF, or post-essential thrombocythemia MF, according to the 2008 revised World Health Organization criteria
* Intermediate-1, intermediate-2, or high-risk according to the IWG-MRT Dynamic International Prognostic Scoring System
* Life expectancy >= 6 months
* Peripheral blood blast count of less than (<) 10%
* Palpable splenomegaly of greater than (>) 5 centimeters (cm) below the left costal margin
* Eastern Cooperative Oncology Group performance status of 0 to 2
* Adequate hepatic and renal function

Exclusion Criteria:

* Prior treatment with a Hedgehog or Janus kinase pathway inhibitor
* Treatment with strong cytochrome P450 3A4 inhibitors/inducers within 28 days prior to Day 1
* Prior therapy for the treatment of intermediate- or high-risk MF including chemotherapy, interferon, thalidomide, busulfan, lenalidomide, anagrelide, or androgens within 28 days prior to Day 1
* Prior splenectomy or splenic irradiation
* Inadequate bone marrow reserve
* Participants with any history of platelet counts of < 50,000/mccL or ANC of < 500/mL, except during treatment for myeloproliferative neoplasm or treatment with cytotoxic therapy for any other reason
* Planned allogeneic bone marrow transplant during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-01-25 (Actual); Primary Completion 2017-03-29 (Actual); Study Completion 2017-07-12 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants who Achieve a Greater Than or Equal to (>=) 35% Reduction in Spleen Volume from Baseline at Week 24 | Week 24
  Determined by an Independent Review Committee (IRC) Using International Working Group-Myeloproliferative Neoplasms Research and Treatment (IWG-MRT) Revised Response Criteria
Percentage of Participants with Complete Remission (CR) and Partial Remission (PR) at Week 24, as Determined by an IRC Using IWG-MRT Revised Response Criteria | Week 24

SECONDARY OUTCOMES:
Plasma Vismodegib Concentration at Steady State | Predose (0 hour) on Weeks 6, 12, 24, 36, and 48
Unbound Vismodegib Concentration at Steady State | Predose (0 hour) on Weeks 6, 12, 24, 36, and 48
Alpha 1-Acid Glycoprotein Concentration at Steady State | Predose (0 hour) on Weeks 6, 12, 24, 36, and 48
Percentage of Participants who Achieve a >= 35% Reduction in Spleen Volume from Baseline, as Determined by an IRC Using IWG-MRT Revised Response Criteria at Week 48 | Baseline, Week 48
Percentage of Participants who Achieve a >= 35% Reduction in Spleen Volume from Baseline, as Determined by an Investigator at Weeks 24 and 48 | Baseline, Weeks 24 and 48
Percentage of Participants with CR and PR, as Determined by an IRC Using IWG-MRT Revised Response Criteria at Week 48 | Week 48
Percentage of Participants with CR and PR, as Determined by an Investigator at Weeks 24 and 48 | Weeks 24 and 48
Percentage of Participants with Overall Response Rate (CR, PR, and Clinical Improvement) at Weeks 24 and 48, as Determined by an IRC Using IWG-MRT Revised Response Criteria | Weeks 24 and 48
Percentage of Participants with Overall Response Rate (CR, PR, and Clinical Improvement) at Weeks 24 and 48, as Determined by the Investigator Using IWG-MRT Revised Response Criteria | Weeks 24 and 48
Percentage of Participants who Achieve Anemia Response at Weeks 24 and 48, as Determined by the Investigator Using IWG-MRT Revised Response Criteria | Weeks 24 and 48
Percentage of Participants with Symptom Response (Participants who Achieve a >= 50% Reduction from Baseline in the Myeloproliferative Neoplasm Symptom Assessment Form [MPN-SAF] Total Symptom Score [TSS]) | Baseline, Weeks 24 and 48
Duration of Response, as Determined by the Investigator and an IRC Using IWG-MRT Revised Response Criteria or Death from Any Cause During the Study | Baseline up to 28 days after the last dose of study drug (52 weeks)
Percentage of Participants with Improvement from Baseline in Bone Marrow Fibrosis at Weeks 24 and 48, as Determined by the Investigator Using the European Consensus Grading System | Baseline, Weeks 24 and 48
Percentage of Participants with Improvement from Baseline in Bone Marrow Fibrosis at Weeks 24 and 48, as Determined by Independent Pathology Review Using the European Consensus Grading System | Baseline, Weeks 24 and 48
Progression-Free Survival | Baseline up to the end of the study (up to 1 year after completing 48 weeks of treatment by the last participant)
Percentage of Participants who Achieve a >= 50% Reduction in Fatigue from Baseline to Weeks 24 and 48 as Measured by MPN-SAF TSS | Baseline, Weeks 24 and 48
Percentage of Participants who Achieve a >= 50% Reduction in Other Symptom and Impact Item Scores from Baseline to Weeks 24 and 48, as Measured by the MPN-SAF | Baseline, Weeks 24 and 48
Percentage of Participants who Achieve a Meaningful Improvement on the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 Scale Scores from Baseline to Weeks 24 and 48 | Baseline, Weeks 24 and 48
  Meaningful improvement is defined as a 10-point change.
Overall Survival | Baseline up to the end of the study (up to 1 year after completing 48 weeks treatment by the last participant)
Percentage of Participants with Adverse Events (AEs) | Baseline up to Month 48

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (13):
- United States (6):
  - Florida Cancer Specialists-Broadway, Fort Myers, Fort Myers, Florida
  - Florida Cancer Specialist, North Region, St. Petersburg, Florida
  - Florida Cancer Specialists, West Palm Beach, Florida
  - Oncology Hematology Care Inc, Cincinnati, Ohio
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Uni of Texas - Md Anderson Cancer Center; Dept of Leukemia, Houston, Texas
- Canada (3):
  - Tom Baker Cancer Centre-Calgary; Clinical Research Unit, Calgary, Alberta
  - Queen Elizabeth II Health Sciences Centre; Oncology, Halifax, Nova Scotia
  - Centre Hospitalier De L'Universite De Montreal, Hopital Notre-Dame, Montreal, Quebec
- Germany (2):
  - Uniklinik RWTH Aachen; Med. Klinik IV; Klinik für Hämatologie, Onkologie, Hämostaseologie und Stammz, Aachen
  - Campus Virchow-Klinikum Charité Centrum 14; Medizinische Klinik m.S. Hämatologie u. Onkologie, Berlin
- Italy (2):
  - A.O.U. Citta' Della Salute E Della Scienza-P.O. Molinette;S.C. Ematologia, Turin, Piedmont
  - Az. Osp. Di Careggi; Divisione Di Ematologia, Florence, Tuscany

REFERENCES:
- [Derived] Couban S, Benevolo G, Donnellan W, Cultrera J, Koschmieder S, Verstovsek S, Hooper G, Hertig C, Tandon M, Dimier N, Malhi V, Passamonti F. A phase Ib study to assess the efficacy and safety of vismodegib in combination with ruxolitinib in patients with intermediate- or high-risk myelofibrosis. J Hematol Oncol. 2018 Sep 24;11(1):122. doi: 10.1186/s13045-018-0661-x. PMID 30249277